CLINICAL TRIAL: NCT03016676
Title: Study of Spinal Manipulation(SM) Decrease Postural Instability and Improve Quality of Life in Patients With Chronic Non Specific Low Back Pain
Brief Title: Efficacy of SM on Postural Instability and Quality of Life in Patients With Chronic Non Specific Low Back Pain(CNSLBP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lovely Professional University (Other)
Responsible Party: Principal Investigator, Kanchan Sarker, PhD Research Scholar, Lovely Professional University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LPU-11304873
Record Dates: First submitted 2016-12-31; First posted 2017-01-10 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Non Specific Low Back Pain
Keywords: Spinal Manipulation; Postural Instability; Quality of Life
MeSH Terms: interventions — Manipulation, Spinal; Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spinal manipulation (Experimental): Spinal manipulation -High velocity low amplitude thrust (HVLA), Dosages : 2 repetition at the same time, Duration-10-20 minutes. total 2 weeks.
  Interventions: Other: Spinal Manipulation
- Exercise therapy (Experimental): Exercise Therapy(ET): Exercise therapy (ET) 3 program: self education, supervised exercise visits, and home exercise. Duration-45 minutes,Total number of visits 12 for 2 weeks.
  Interventions: Other: Exercise therapy

INTERVENTIONS:
Other: Spinal Manipulation — High velocity low amplitude thrust (HVLA) to the lumbar region of the spine between L1 and L5 vertebrae. The exact level thrust will be at the discretion of the treating practitioner determined by the level with the greatest perceivable motion restriction. The HVLA thrust will be performed with the patient side lying in a neutral.They take part in 12 treatment visits, 10 to 20 minutes sessions of SM over 2 weeks. Light soft tissue techniques (i.e., active and passive muscle stretching, and ischemic compression of tender points) may be used as needed to facilitate the manual therapy.
  Arms: Spinal manipulation
Other: Exercise therapy — Self education, supervised exercise visits, and home exercise. The overall objectives are to help patient's mange their LBP and prevent future LBP recurrences. Total number of visits 12.Each visit starts with 10 minutes of self-care education to help patients establish and monitor goals aligned with the exercise program and enhance their understanding of LBP. Participants will be taught the importance of movement and activity, pain management techniques, and methods for developing spinal posture awareness during activities of daily living (e.g., lifting, pushing, pulling, sitting, getting out of bed, and using a backpack).
  Arms: Exercise therapy

SUMMARY:
This study will give a new insight to the physiotherapy fraternity in the effects of spinal manipulation in as clinical practice, as well as the patient's community in quick re-establishment of functional ability, pain decrease, and improvement of quality of life for economic reasons. In this high opinion, application of short-term intensive spinal manipulation for non specific chronic low back pain treatment is desirable.

DETAILED DESCRIPTION:
The protocol for group A included High velocity low amplitude thrust (HVLA) to the lumbar region of the spine between L1 and L5 vertebrae.The HVLA thrust will be performed with the patient side lying in a neutral.52 They take part in 12 treatment visits, 10 to 20 minutes sessions of SM over 2 weeks. Light soft tissue techniques (i.e., active and passive muscle stretching, and ischemic compression of tender points) may be used as needed to facilitate the manual therapy.

The protocol for group B included sets of exercise therapy. There are three components to the exercise therapy (ET) program: self education, supervised exercise visits, and home exercise. The overall objectives are to help patient's manage their LBP and prevent future LBP recurrences. Total number of visits 12 (e.g., ability to perform exercises independently).

Outcome:

Patient self-report outcomes will be collected at first baseline visit and its base on the pain intensity and quality of life will be assessed by using numerical pain rating scale and EuroQol questionnaire. Objective outcome measures will be collected at the first baseline visit and its base on postural instability and pressure pain threshold will be assessed by using Win track platform and digital algometer.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 55 years of age.
* Both genders.
* Subjects diagnosed with non-specific chronic low back pain with duration of >3 months.
* Low back pain intensity≥3 on 0-10 in numerical pain rating scale.

Exclusion Criteria:

* Injury or surgery of spine.
* Congenital spinal deformity (e.g Spina bifida, Scoliosis, ankylosing spondylitis etc )
* Lumbar radiculopathy or presenting neurological deficit.
* Subjects administered Epidural injection.
* Contra-indication to manipulations-vertebral malignancy, vertebral-basilar insufficiency, bone infections, fracture.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2015-07; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Patients with CNSLBP will received SM and ET to measure postural instability to assess after 12 session over 2 weeks. | Baseline before treatment and after 2 week of treatment
  Clinical outcomes will be assessed at baseline and following 2 weeks of participation in the study,Change from baseline in postural instability will be measured by Win Track Platform at 2 weeks.
Patients with CNSLBP will be received SM and ET to measure quality of life to assess after 12 session over 2 weeks. | Baseline before treatment and after 2 week of treatment
  Clinical outcomes will be assessed at baseline and following 2 weeks of participation in the study, Change from baseline in quality of life on EuroQoL questionnaire at 2 weeks.EuroQol questionnaire is a wide accepted questionnaire for health-related quality of life and consists of two components. Its first component (EQ-5D-5L) consists of five dimensions (mobility, self-care, usual activity, pain/discomfort, and anxiety/depression). However, each dimension now has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems.
Patients with CNSLBP will be received SM and ET to measure Pain intensity to assess after 12 session over 2 weeks. | Baseline before treatment and after 2 week of treatment
  Clinical outcomes will be assessed at baseline and following 2 weeks of participation in the study, Change from baseline in pain instability on Numerical pain rating scale (NPRS). An11-point numeric pain rating scale will be used to assess pain intensity (primary outcome measure), with 0 representing "no pain" and 10 representing the "worst possible pain" at the time of the assessment. Pain intensity will be measured before and after treatment.
Patients with CNSLBP will be received SM and ET to measure Pain sensitivity(Pressure pain threshold-PPT) to assess after 12 session over 2 weeks. | Baseline before treatment and treatment after 2 week of treatment
  Clinical outcomes will be assessed at baseline and following 2 weeks of participation in the study, Change from baseline in pain sensitivity (PPT) on Digital algometer.Pain sensitivity (PPT) will be measured on the lumbar area bilaterally. Digital Algometer (Jagson scientific Industries, Ambala-133001, Haryana, India) will be used with a circular rounded aluminium tip, 1 cm2, and with an application rate of 25 KN/s. The measurements will be performed twice and the average of the two registrations will be filed.

CONTACTS AND LOCATIONS:
Overall Officials: Kanchan Ku Sarker, Ph.D, Principal Investigator — Lovely Professional University,Phagwara, Kapurthala, Punjab, India.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Kanchan Sarker, U K Mohanty, Jasobanta Sethi, <em><a href="http://citeweb.info/20160278206">EFFECT OF SPINAL MANIPULATION ON POSTURAL INSTABILITY IN PATIENTS WITH NON SPECIFIC LOW BACK PAIN</a></em> (2016) — http://www.ijpbs.net/abstract.php?article=5240
- Available data/document: Study Protocol — http://www.ijpbs.net/abstract.php?article=5240